CLINICAL TRIAL: NCT01782183
Title: Thermographic Characteristics of Sore Throat by Thermographic Camera
Acronym: thermography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Doron Carmi (Other)
Responsible Party: Sponsor-Investigator, Doron Carmi, Medical Doctor, Clalit Health Services
Organization: Clalit Health Services (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: COM120017CTIL
Record Dates: First submitted 2013-01-01; First posted 2013-02-01 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Fever; Sore Throat
Keywords: sore throat; thermal camera photo; normal tonsils and pharynx; redness of tonsils and/or pharynx; exudates on tonsils; petechiae of the palate
MeSH Terms: conditions — Fever; Pharyngitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thermal camera by Flir HM series (Experimental): all patients in both study and control groups will undergo thermal camera photo of the tonsils by Flir HM series
  Interventions: Device: Thermal camera by Flir -HM series.

INTERVENTIONS:
Device: Thermal camera by Flir -HM series. — The patient will be photographed twice by directing the camera externally to each tonsil from below the mandibular angle

SUMMARY:
Thermographic cameras are used to determine temperature and temperature differences. Attempts have been made to use the thermographic camera as a diagnostic tool in clinical practice. Thermographic cameras have been approved by the FDA in the diagnosis of breast cancer. The camera absorbs infrared radiation which is discharged from the tissue and than translates it to a digital data or a photograph. The camera does not radiate and direct contact with the patient is not needed. The safety is similar to a regular optic camera. No study on thermographic characteristics of inflammation of organs has been published. The purpose of this study is to demonstrate and document these characteristics of inflammation. The correlation between the thermographic imaging and the clinical diagnosis, using routine methods, will be analyzed. The differences of thermographic imaging between an inflamed organ of a subject to a non inflamed same organ of a normal control will also be analyzed. The management of the patient will be by standard practice and will not be influenced by the thermographic camera image and the study outcome.

DETAILED DESCRIPTION:
Patients aged between 5 years and 18 years, who attend the primary health clinic for medical treatment with a complaint of only sore throat and fever will be offered to participate in the study and have a thermal camera photo of the tonsils. The study group will consist of 100 patients. Fifty patients will be enrolled who present with sore throat and another 50 patients will be enrolled who present to the clinic for any febrile condition other than a sore throat. A parent will sign consent after the parent and child have received an explanation about the study. The patient will be photographed twice by directing the camera externally to each tonsil from below the mandibular angle. The photograph will be saved in the camera and the investigator will not be able to see the photo. The number of the photograph will be listed with the patient name. The investigator will keep the list and only he will have access to the clinical data. Thereafter a standard clinical examination will be performed and all the patients will receive standard medical treatment irrespective of their participation in the study. The description of the tonsils and the pharynx will be recorded in the patient's electronic medical file and will consist of the following information (one or more of the following options): normal tonsils and pharynx, redness of tonsils and/or pharynx, exudates on tonsils, petechiae of the palate. Patients who will not have the full description as described above will be excluded from analysis from the study. The data will be analyzed descriptively for a correlation between the clinical findings and the thermal photograph

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 5 years and 18 years who attend the primary health clinic for medical treatment with a complaint of sore throat and fever
2. The control group will consist of patients with fever aged between 5 years and 18 years who attend the primary health clinic for medical treatment complaint other than sore throat

Exclusion Criteria:

1. Patients who are already treated with antibiotics

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between the symptoms of sore throat and fever and the temperature of the tonsils as measured by the thermal photograph. | one day

SECONDARY OUTCOMES:
Correlation between clinical diagnosis of tonsillitis and thermal camera photo | one day
  Correlation between tonsillitis characterized by redness of tonsils and/or pharynx, exudates on tonsils, petechiae of the palate and temperature of the tonsils as measured by the thermal camera photo.

CONTACTS AND LOCATIONS:
Overall Officials: Doron Carmi, MD, Principal Investigator — Clalit Health Services
Locations (1):
- Primary Care Clinic of Clalit Health Services, Tel Aviv, Israel